CLINICAL TRIAL: NCT06487468
Title: A Study on Risk Factors in Heart Failure Patients With Preserved Ejection Fraction After Hospital Discharge
Brief Title: Risk Factors In Heart Failure Patients With Preserved Ejection Fraction
Acronym: RIPE-HF
Status: Completed | Type: Observational
Sponsor: Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Jianping Zeng, Director of Cardiovascular Department of Xiangtan Central Hospital,Clinical Professor, Xiangtan Central Hospital
Other Study IDs: 2024/6
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF, Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFpEF Group: HFpEF (Heart failure with preserved ejection fraction): LVEF≥50%.
  Non-endpoint events group versus Endpoint events (all-cause death,cardiovascular death or heart failure readmission) group

SUMMARY:
This study aimed to identify the independent risk factors associated with heart failure readmission, cardiac mortality and all-cause death among patients discharged from Xiangtan Central Hospital with heart failure and preserved ejection fraction (HFpEF). Understanding related risk factors might add future clinical decision making for individualized post discharge management of HFpEF patients aiming to improve the outcome of discharged HFpEF patients.

DETAILED DESCRIPTION:
This study sought to determine the independent risk factors linked to endpoint events (which include all-cause mortality or readmission for heart failure, cardiovascular death) among hospitalized patients with heart failure and preserved ejection fraction (HFpEF) at Xiangtan Central Hospital during the period from May 1, 2014, to January 31, 2023. The clinical follow up ended on January 31, 2024. The study examined the risk factors associated with the endpoint outcome (cardiovascular death and death from any cause and readmission due to heart failure) to provide clinical evidence for intervening discharged HFpEF patients, with the objective of improving patient outcomes in future clinical practice.

The clinical features of hospitalized heart failure with preserved ejection fraction (HFpEF, EF≥50%) are analyzed retrospectively by reviewing the patient's demographic, clinical data, including patient medical history, initial clinical evaluations, and therapeutic interventions, as well as echocardiographic data in the hospital's electronic health records and relevant databases. The clinical outcome of enrolled patients are obtained through a team of three experienced cardiologists and twelve nursing professionals through outpatient consultations, telephone follow-ups, and community visit. The primary endpoint events are all-cause mortality, the second endpoints are the composite cardiovascular death and heart failure readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged with diagnosis of heart failure were screened and met definition of heart failure with preserved ejection fraction (HFpEF) according to the 2021 European Society of Cardiology (ESC) guidelines at final analysis.
* 1）Heart failure signs and symptoms; 2）LVEF>50%;

Exclusion Criteria:

* 1) age under 18 years; 2) life expectancy of less than one year due to non-cardiac conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who hospitalized the Xiangtan Central Hospital between May 1, 2014, and January 31, 2023, with the diagnosis of heart failure and met HFpEF criteria at final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 9419 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
All-cause death（people） | The patients are clinically followed up until January 31, 2024, per clinical visit or telephone call or community visit.
  Risk factors of all-cause death are analyzed（Increase the factors that contribute to the occurrence of endpoint events）

SECONDARY OUTCOMES:
Cardiovascular death and Heart failure readmission（people） | The patients are clinically followed up until January 31, 2024, per clinical visit or telephone call or community visit.
  The risk factors related to cardiovascular death and heart failure readmission post discharge are analyzed.（Increase the factors that contribute to the occurrence of endpoint events）

REFERENCES:
- [Derived] Zhu Y, Zhao W, Liu Z, Tan D, Tao L, He W, Jiang K, Huang H, Wu M, Tang L, Zeng J, Zhou S. Development and validation of a prediction model for all-cause death in heart failure patients with preserved ejection fraction: a single-centre cohort study in China. BMJ Open. 2025 Sep 10;15(9):e094909. doi: 10.1136/bmjopen-2024-094909. PMID 40935414